CLINICAL TRIAL: NCT05309876
Title: Secondary Prevention of Cardiovascular Disease With the Lifestyle Tool
Brief Title: Secondary Prevention With the Lifestyle Tool
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lifestyle3
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants get access to the tool or get assigned to a control group without access
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usage of tool (Experimental): Participants get access to the tool and use it regularly
  Interventions: Behavioral: Lifestyle tool
- Controls on usual care (No Intervention): Participants who get randomized to control cannot access the tool. Development of cardiovascular disease is followed via clinical registries.

INTERVENTIONS:
Behavioral: Lifestyle tool — Regular use of the digital Lifestyle tool
  Arms: Usage of tool

SUMMARY:
In this study participants will be randomized to use a digital lifestyle tool over three years or to a control group without access to the tool. The investigators will prospectively follow the incidence of major cardiovascular events in patients who have previously suffered from a myocardial infarction in those using the tool regularly and those in the control group.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains a leading cause of death in most European countries, and new strategies for prevention are urgently needed.

Previous studies on primary and secondary prevention have shown that lifestyle interventions can affect risk factors for CVD and reduce cardiovascular morbidity and mortality. Many prevention programmes are, however, time-limited and fail to provide continuous support. They also require substantial costs and healthcare resources. Furthermore, accessibility to primary and secondary cardiac prevention programmes is highly variable, as is long-term adherence to lifestyle advice.

In light of this, international associations have emphasized the need for innovative, scalable and cost-effective lifestyle interventions that could be integrated into pre-existing healthcare structures. Digital tools have large potential for clinical utility, but there are several important knowledge gaps. First, data on long-term efficacy is scarce. Second, most studies to date have included only small number of individuals, and there is a need for large randomized controlled studies. Third, cost-effectiveness remains to be demonstrated.

The objective or this study is to evaluate a new web-based tool, developed at the University Gothenburg, Sweden, that aims to support patient autonomy and motivation to make sustainable lifestyle changes.

In individuals who have previously suffered from a myocardial infarction the investigators will test the hypothesis that those who access to the tool have lower incidence of further major cardiovascular events (MACE) compared with control individuals.

The study is an investigator-initiated single-center study conducted over three years.

The tool is web-based and used via a computer or mobile phone. It is used at each individual's preferred pace but participants are recommended to login at least every other week. Every round the participants choose a themes (out of appr. 80 possible covering e.g. food, exercise, stress, self-reflection aspects), which takes appr. 15-30 minutes to complete. Participants then reflect on the content and how it could be implemented in daily life. When returning for next round participants are asked to reflect on any changes done since last time.

ELIGIBILITY:
Inclusion Criteria:

* age 35 to 80 years
* myocardial infarction within one year prior to enrolment
* access to computer or mobile phone.

Exclusion Criteria:

* conditions or treatments that in the judgement of the Investigator could affect the study evaluation

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11000 (Estimated)
Dates: Start 2022-04-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse cardiovascular event | 3 years
  Incidence of major adverse cardiovascular event, defined as cardiovascular death, myocardial infarction, stroke, or hospitalization for heart failure compared between participants regularly using the tool and on usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Rosengren, Professor, Principal Investigator — Göteborg University
Locations (1):
- Skane University Hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results will be shared after deidentification.
Time Frame: Data will be available after publication.
Access Criteria: To researchers who provide a methodologically sound proposal in order to achieve the aims of that proposal. Proposals should be directed by email to internetverktyg@gu.se